CLINICAL TRIAL: NCT05480280
Title: mFOLFOX6 Combined With Dalpiciclib(SHR6390) in Patients With Metastatic Colorectal Cancer (FIND): A Single-arm, Phase IIa Study.
Brief Title: mFOLFOX6 Combined With Dalpiciclib in Patients With Metastatic Colorectal Cancer
Acronym: FIND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaojian Wu, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-057
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Advanced/Metastatic Colorectal Cancer
Keywords: Colorectal cancer, Dalpiciclib, Efficacy and safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — dalpiciclib; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This is an prospective, single-center, single-arm, Simon's two-stage design, phase IIa study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFOX6 + dalpiciclib (Experimental): Dalpiciclib is orally administered at 125mg qd for 21 days and discontinue for 7 days. mFOLFOX6 will be administered every 2 weeks.
  Interventions: Drug: Dalpiciclib; Drug: Oxaliplatin injection; Drug: Calcium folinate; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib is orally administered at 125mg qd for 21 days and discontinue for 7 days.
  Other Names: SHR6390
Drug: Oxaliplatin injection — 85mg/m², ivdrip, D1
  Other Names: L-OHP
Drug: Calcium folinate — 400mg/m², ivdrip, D1; or calcium levofolinate, 200 mg/m², ivdrip, D1
  Other Names: Leucovorin
Drug: 5-fluorouracil — 400mg/m², iv, D1; and 2400mg/m², civ, 46-48h
  Other Names: Fluorouracil; 5-FU

SUMMARY:
This is an prospective, single-center, single-arm, Simon's two-stage design, phase IIa study for advanced/metastatic colorectal cancer (CRC) who had failed or were intolerant to standard treatment. This study aims to evaluate the safety and efficacy of mFOLFOX6 combined with dalpiciclib (SHR6390) in the treatment of advanced/metastatic colorectal cancer.

DETAILED DESCRIPTION:
1. Primary study end point:

   To evaluate the safety and objective response rate (ORR) of mFOLFOX6 combined with dalpiciclib (SHR6390) in patients with advanced/metastatic colorectal cancer who had failed or were intolerant to standard treatment.
2. Secondary study end Point:

To evaluate the progression-free survival (PFS) and overall survival (OS) of mFOLFOX6 combined with dalpiciclib (SHR6390) in patients with advanced/metastatic colorectal cancer who had failed or were intolerant to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign informed consent
* Age: from 18 to 70 years old
* Definite histological evidence of colorectal adenocarcinoma
* ECOG 0-1
* Advanced or metastatic colorectal cancer (AJCC/UICC stage IV) is confirmed by enhanced CT of the chest, abdomen and pelvis, with evaluable lesions
* Tumor progression or intolerable toxicity after previous standard treatment; Tumor progression during adjuvant therapy or within 6 months after completion of adjuvant therapy was considered as first-line treatment (Standard treatment must include all of the following drugs: fluorouracil, irinotecan, and oxaliplatin; With or without anti-VEGF monoclonal antibody (bevacizumab); Anti-EGFR treatment(cetuximab or panitumumab) in left colorectal RAS (KRAS/NRAS) wild-type subjects)
* The bone marrow, liver and kidney function satisfies the following conditions within 7 days before treatment (including day 7):

Hemoglobin ≥90g/L, neutrophil count ≥1.5×109/L, platelet count ≥75×109/L; aspartate aminotransferase (AST) ≤ 2 upper limit of normal (ULN), glutaminate alanine transaminase (ALT) ≤ 3 ULN, total bilirubin ≤ 1.5 ULN, serum creatinine ≤ 1.5 ULN

* Peripheral neurological lesions recover (≤ grade 1) before enrollment
* Subjects should not participate in other clinical trials during the study period
* Willing and able to comply with research procedures and follow-up plan

Exclusion Criteria:

* Complicated with obstruction, active bleeding or perforation and requiring emergency surgery or stent placement
* Existing or coexisting other active malignancies
* Previously CDK inhibitors treatment
* Major surgery or severe trauma such as laparotomy, thoracotomy or laparoscopic organ removal within the previous 4 weeks
* Active coronary artery disease, severe/unstable angina or newly diagnosed angina or myocardial infarction in the past 12 months
* Thrombotic or embolic events occurred within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism or deep vein thrombosis
* New York Heart Association (NYHA) Class II or higher Congestive heart failure
* Presence of clinically symptomatic third space effusion (eg, massive pleural or ascites) that cannot be controlled by drainage or other methods
* Human immunodeficiency virus (HIV) infection or diseases associated with acquired immunodeficiency syndrome (AIDS)
* Active inflammatory bowel disease or other colorectal disease leading to chronic diarrhea
* Presence of CTCAE grade 2 or higher toxicity (other than anemia, alopecia and skin pigmentation) that has not recover due to any previous treatment
* Suspected allergies to any of the relevant drugs used in the study
* Pregnant or lactating
* Women of childbearing age (<2 years after last menstrual period) or men of childbearing potential not using or refusing to use effective non-hormonal contraception
* Any unstable medical condition that affects patient safety and study compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Adverse Events) | 1 year
  The number of subjects who had adverse events and the type of adverse events were recorded according to CTCAE V.5.0. Safety failure was defined as any grade 3-5 treat-related adverse event (AE) (CTCAE 5.0) within 90 days from the date of the last regimen (whichever was reached later).
Objective Response Rate (ORR) | 1 year
  ORR was defined as the proportion of all subjects who received the study treatment and whose best overall response (BOR) was a complete response (CR) or a partial response (PR) according to RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 1 year
  PFS was defined as the date from enrollment to the first recorded of tumor progression (assessed by RECIST version 1.1) or the date of death from any cause, whichever came first.
Overall Survival (OS) | 1 year
  OS was defined as the date from enrollment to the date of death or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojian Wu, Ph.D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No